CLINICAL TRIAL: NCT03674320
Title: Cycled Testosterone Administration During Pulmonary Rehabilitation in Early Stage COPD
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: No Funding
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-0202
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2021-01

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — testosterone enanthate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo (saline) injections will be given via intramuscular injection at study weeks 2,3, 6, 7, 10, and 11.
  Interventions: Drug: Placebo
- Testosterone Enanthate (Active Comparator): Testosterone Enanthate (100mg men, 25mg women) will be given via intramuscular injection at study weeks 2, 3, 6, 7, 10 and 11.
  Interventions: Drug: Testosterone Enanthate

INTERVENTIONS:
Drug: Testosterone Enanthate — Testosterone Enanthate (25 mg women, 100mg men) will be given via intramuscular injection at study week 2, 3, 6, 7, 10 and 11.
  Arms: Testosterone Enanthate
Drug: Placebo — Placebo Injection (saline) will be given via intramuscular injection at study week 2, 3, 6, 7, 10 and 11.
  Arms: Placebo

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is characterized by chronic inflammation of the airways and/or damage to the lungs which leads to progressive impairment in airflow and the ability to breathe. COPD affects 6 to 20% of the US population and is among the leading causes for mortality in men and women. While COPD is principally a pathology of the airway, skeletal muscle wasting is a widely recognized comorbidity contributing to frequent and expensive hospital visits.

Hospital readmission rates among COPD patients are high and the majority of the readmissions are considered preventable. The reasons COPD patients lose muscle are still poorly understood although reduced pulmonary function has been associated with reduced testosterone levels. Muscle building treatments, including testosterone therapy, with and without exercise, have consistently been shown to promote improvements in body composition, exercise capacity, and health related quality of life of COPD patients.

The overall goal of this investigation is to provide an effective long-term treatment strategy that prevents the advancement of COPD in men and women through a safe, cycled administration of testosterone during the early stages of disease.

DETAILED DESCRIPTION:
Male and female COPD patients participating in a 12 week pulmonary rehabilitation program at the University of Texas Medical Branch enrolled in the study will be randomized into either placebo or testosterone enanthate (100mg men, 25mg women) treatment. Testosterone and placebo will be given in a cyclic fashion during the pulmonary rehabilitation with single injections given on weeks 2, 3, 6, 7, 10 and 11. Baseline (during week 1 of rehabilitation) and post (during week 12 of rehabilitation) study testing will measure the effectiveness of testosterone on several measures listed in the outcome section.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 40 - 80 years
2. Stable weight (<10 lbs change in past 12 months - self reported)
3. (Willing to) participate in pulmonary rehabilitation (PR) program at UTMB
4. Air flow limitation based on spirometry (FEV1 < 60% predicted) (prior to PR)
5. Daily symptoms according to COPD assessment test (CAT) > 15 (prior to PR)

Exclusion Criteria:

1. Late stage COPD, GOLD Stage 3-4 (FEV1 > 60% predicted)
2. Inability to perform 6-minute walking test or other physical therapy activities
3. Inability/unwillingness to follow the pulmonary rehabilitation program
4. Already more than 2 weeks into the pulmonary rehabilitation program at time of consenting
5. Uncontrolled endocrine or metabolic disease (e.g. liver disease, renal disease, diabetes)
6. Uncontrolled hypertension. Systolic blood pressure greater than or equal to 160mm Hg or a diastolic blood Pressure greater than or equal to 100mm Hg on three consecutive measurements taken at one-week intervals. Testosterone can cause fluid retention that could worsen uncontrolled hypertension. Subjects will be included if they are on two or less blood pressure medications and have a blood pressure below these criteria
7. History of angina that occurs with exertion or at rest or a myocardial infarction within the last 12 months
8. LDL cholesterol greater than 200 mg/dL as testosterone administration may elevate LDL cholesterol levels 9. Hematocrit greater than 51%

10. Current use of or history of recent anabolic steroid use (within 3 months) 11. Current abuse of alcohol or recreational drugs 12. Any other condition or event considered exclusionary by the PIs and covering faculty physician 13. Vulnerable populations including: individuals unable to consent on their own behalf, prisoners and pregnant women

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
90 day re-hospitalization rate | 90 days
  Re-hospitalization rates will be collected from the electronic medical record and/or subject interviews.
Exercise Capacity as measured by distanced walked during 6 minute walk test at baseline study testing | baseline
  Exercise capacity will be measured by distance walked in 6 minutes on a predefined course. Subjects will be asked to walk at 100% effort (as quickly as they can safely walk without running) for 6 minutes. Distance traveled for the 6 minutes will be recorded. The walking test will be completed at baseline. Data will be reported as meters (m) walked in 6 minutes.
Exercise Capacity as measured by distanced walked during 6 minute walk test at 12 weeks. | 12 weeks
  Exercise capacity will be measured by distance walked in 6 minutes on a predefined course. Subjects will be asked to walk at 100% effort (as quickly as they can safely walk without running) for 6 minutes. Distance traveled for the 6 minutes will be recorded. The walking test will be completed at baseline. Data will be reported as meters (m) walked in 6 minutes.

SECONDARY OUTCOMES:
Handgrip strength as measured by hand dyanometer at baseline study testing | baseline
  Handgrip strength as measured by hand dyanometer at baseline of pulmonary rehabilatation and study drug intervention. Data will be reported as maximum force produced in kilograms.
Handgrip strength as measured by hand dyanometer at 12 weeks | 12 weeks
  Handgrip strength as measured by hand dyanometer after 12 weeks of pulmonary rehabilatation and study drug intervention. Data will be reported as maximum force produced in kilograms.
Difficulty breathing during the Exercise Capacity Test as measured using the Borg Dyspnea Scale (BDS) at baseline | baseline
  The BDS assesses difficulty breathing during the 6 minute walk test. Patients indicate their level of difficulty on a scale of 0 (no difficult) to 10 (maximal difficulty).
Difficulty breathing during the Exercise Capacity Test as measured using the Borg Dyspnea Scale (BDS) at 12 weeks | 12 weeks
  The BDS assesses difficulty breathing during the 6 minute walk test. Patients indicate their level of difficulty on a scale of 0 (no difficult) to 10 (maximal difficulty).
Lung function as measured by Forced Expiratory Volume (FEV1) at baseline study testing | baseline
  Lung function as measured by Forced Expiratory Volume (FEV1). FEV1 measured the amount of air that can be forcefully exhaled in one second. FEV1 is measured using a standard spirometer. Data will be reported as L of air expelled.
Lung function as measured by Forced Expiratory Volume (FEV1) at 12 weeks | 12 weeks
  Lung function as measured by Forced Expiratory Volume (FEV1). FEV1 measured the amount of air that can be forcefully exhaled in one second. FEV1 is measured using a standard spirometer. Data will be reported as L of air expelled.
Lung Function as measured by Vital Capacity (VC) at baseline | baseline
  Lung function as measured by Vital Capacity (VC) at baseline. VC measures the maximum amount of air that can be exhaled from the lung. VC is measured using a standard spirometer. Data will be reported as L of air expelled.
Lung Function as measured by Vital Capacity (VC) at 12 weeks | 12 weeks
  Lung function as measured by Vital Capacity (VC) at 12 weeks. VC measures the maximum amount of air that can be exhaled from the lung. VC is measured using a standard spirometer. Data will be reported as L of air expelled.
Lung Function as measured by Forced Vital Capacity (FVC) at baseline | baseline
  Lung function as measured by Forced Vital Capacity (FVC) at baseline. FVC measures the maximum amount of air that can be forcibly exhaled from the lungs after taking the deepest breath possible. FVC is measured using a standard spirometer. Data will be reported as L of air expelled.
Lung Function as measured by Forced Vital Capacity (FVC) at 12 weeks. | 12 weeks
  Lung function as measured by Forced Vital Capacity (FVC) at baseline. FVC measures the maximum amount of air that can be forcibly exhaled from the lungs after taking the deepest breath possible. FVC is measured using a standard spirometer. Data will be reported as L of air expelled.
Lung Function as measured by Forced Expiratory Flow 25%-75% Forced Vital Capacity (FEF 25-75) at baseline. | baseline
  Lung Function as measured by Forced Expiratory Flow 25%-75% Forced Vital Capacity (FEF 25-75) at baseline. FEF 25-75 measures the flow (speed) of air coming out of the lung during the middle portion of the forced expiration. FEF 25-75 is measured using a standard spirometer. Data will be reported as L/second.
Lung Function as measured by Forced Expiratory Flow 25%-75% Forced Vital Capacity (FEF 25-75) at 12 weeks. | 12 weeks
  Lung Function as measured by Forced Expiratory Flow 25%-75% Forced Vital Capacity (FEF 25-75) at 12 weeks. FEF 25-75 measures the flow (speed) of air coming out of the lung during the middle portion of the forced expiration. FEF 25-75 is measured using a standard spirometer. Data will be reported as L/second.
Lung Function as measured by Maximal Voluntary Ventilation (MVV)at baseline. | baseline
  Lung Function as measured by Maximal Voluntary Ventilation (MVV) at baseline. MVV measures the maximum volume of air that can be breathed in 15 seconds. MVV is measured using a standard spirometer. Data will be reported as L of air.
Lung Function as measured by Maximal Voluntary Ventilation (MVV)at 12 weeks. | 12 weeks
  Lung Function as measured by Maximal Voluntary Ventilation (MVV) at 12 weeks. MVV measures the maximum volume of air that can be breathed in 15 seconds. MVV is measured using a standard spirometer. Data will be reported as L of air.
Fatigue as measured by Multidimensional Fatigue Symptom Inventory (MFSI) at baseline study testing. | baseline
  Fatigue symptoms will be measured using the 30-item Multidimensional Fatigue Symptom Inventory - Short Form, a validated measure that yields one overall score of total fatigue (range -24-96, with higher scores indicating more fatigue) and five subscales (general, physical, emotional, mental, vigor). With the exception of the vigor subscale, higher scores indicate greater fatigue.
Fatigue as measured by Multidimensional Fatigue Symptom Inventory (MFSI) at 12 weeks | 12 weeks
  Fatigue symptoms will be measured using the 30-item Multidimensional Fatigue Symptom Inventory - Short Form, a validated measure that yields one overall score of total fatigue (range -24-96, with higher scores indicating more fatigue) and five subscales (general, physical, emotional, mental, vigor). With the exception of the vigor subscale, higher scores indicate greater fatigue.
Quality of life as measured by St. George's Respiratory Questionnaire (SGRQ) at baseline. | baseline
  The St. George's Respiratory Questionnaire (SGRQ) measures the impact of the disease on overall health, daily life and perceived wellbeing in patients with obstructive airways disease. Scoring is calculated for three components (Symptoms, Activity and Impacts), these components are summed to create a total score. Total scores range from 0 to 100, with higher scores indicating more limitations.
Quality of life as measured by St. George's Respiratory Questionnaire (SGRQ) at 12 weeks. | 12 weeks
  The St. George's Respiratory Questionnaire (SGRQ) measures the impact of the disease on overall health, daily life and perceived wellbeing in patients with obstructive airways disease. Scoring is calculated for three components (Symptoms, Activity and Impacts), these components are summed to create a total score. Total scores range from 0 to 100, with higher scores indicating more limitations.
Quality of Life as measured by COPD Assessment Test (CAT) at baseline study testing | baseline
  The COPD Assessment Test (CAT) is an 8-item questionnaire measuring the impact of COPD on wellbeing and daily life. Each question is rated from 0 (lowest impact) to 5 (highest impact). Scores from each question are summed to calculate a total score. Total scores range from 0 to 40, with higher scores indicating higher impact from COPD. Classification of total score: 0-10 (low impact); 11-20 (medium impact); 21-30 (high impact); 31-40 (very high impact).
Quality of Life as measured by COPD Assessment Test (CAT) at 12 weeks | 12 weeks
  The COPD Assessment Test (CAT) is an 8-item questionnaire measuring the impact of COPD on wellbeing and daily life. Each question is rated from 0 (lowest impact) to 5 (highest impact). Scores from each question are summed to calculate a total score. Total scores range from 0 to 40, with higher scores indicating higher impact from COPD. Classification of total score: 0-10 (low impact); 11-20 (medium impact); 21-30 (high impact); 31-40 (very high impact).
Quality of life as measured by Hospital Anxiety & Depression Scale (HADS) at baseline. | baseline
  The Hospital Anxiety & Depression Scale (HADS) is a 14-item questionnaire with 7 questions measuring anxiety and 7 questions measuring depression. Depression and anxiety will each have their own total score (0-21). Scores classifications: 0-7 (normal); 8-10 (mild); 11-14 (moderate); 15-21 (severe).
Quality of life as measured by Hospital Anxiety & Depression Scale (HADS) at 12 weeks. | 12 weeks
  The Hospital Anxiety & Depression Scale (HADS) is a 14-item questionnaire with 7 questions measuring anxiety and 7 questions measuring depression. Depression and anxiety will each have their own total score (0-21). Scores classifications: 0-7 (normal); 8-10 (mild); 11-14 (moderate); 15-21 (severe).
Total serum testosterone at baseline | baseline
  Total serum testosterone will be measured at baseline by the UTMB Clinical Laboratory.
Total serum testosterone at 12 weeks | 12 weeks
  Total serum testosterone will be measured at baseline by the UTMB Clinical Laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Randall J Urban, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No